

#### Informed Consent Form (ICF) - EXPERT

Researchers: Prof. Dra Eliseth Ribeiro Leão (Advisor) Enfa Lidiane Soares Sodré da Costa (Master Degree Student)

Research title: "Evidence-Based Practice: Proposed Application of Facilitating Tools for Clinical Nurses"

Dear SPECIALIST:

Version 2 - January 2020

We would like to invite you to participate as a volunteer in the research entitled: "Evidence-Based Practice: Proposal for the Application of Facilitator Tools for Clinical Nurses", which refers to the Professional Master's Course Completion Course Teaching in Health. The objectives of this study are:

- 1) Verify the adequacy of the authorized translation of the Portuguese language version of the guide tools of the Johns Hopkins Center for Evidence-Based Practice (Johns Hopkins Center for Evidence-Based Practice), located in the United States.
- 2) Analyze, from the perspective of the clinical nurse, if these tools are facilitators in the structuring and description of an Evidence-Based Practice (EBP) project;
- 3) Analyze, from the researcher's perspective, whether the PBE project met the requirements of: elaboration of a clinical question, bibliographic survey, critical evaluation of the evidence, summary of the evidence and elaboration of the dissemination plan;
- 4) Verify whether previous attitudes and knowledge regarding the implementation of PBE influence the structuring of a PBE project.

|-------------------|--------------------|----------|
| Researcher Rubric | Participant rubric | - |



His form of participation in the study consists of, after evaluating the EBP guide tools in the Portuguese language version of the Johns Hopkins Nursing Evidence-based Practice model (Johns Hopkins model - Evidence-Based Nursing Practice), answering a questionnaire for intelligibility analysis of translation and perform the verification of adequacy with suggestions of the items that need to be addressed or improved, so that we can include the data of your evaluation in this research.

An email will be sent with the original versions in English and the translated versions of each tool into Brazilian Portuguese, as well as the questionnaire with closed questions and suggestions for improvements.

You will not be charged anything and you will not be charged for your participation in this survey.

Regarding the risks of your participation in this research, the form may contain questions that require time for analysis with minimal risk of wear and tear. You can refuse to answer any questions that make you feel uncomfortable. If you have concerns after completing the form, you are encouraged to contact the person responsible for the study. In addition, only researchers will have access to personal information and data. There are no other risks related to your participation in the project.

There are no direct benefits for you if you complete the procedures in this survey. There is a direct benefit expected for professionals who participate in the workshops regarding knowledge in PBE, associated with the possibility of using the tools that you have validated. Future professionals may benefit from what is learned and made available by this study.

We emphasize that your participation in this research is independent of your professional or academic activity at the institution, it is ensured that there will be no type of retaliation if you refuse to participate in this research.


| Researcher Rubric | Participant rubric |
|-------------------|--------------------|

Version 2 - January 2020



## I understand that the following statements about this research are true:

- 1. I can ask any question to the person in charge of the study, Lidiane Soares Sodré da Costa. I can contact you at (11) 99625-3924. I can also contact the institution's Ethics Committee (Research Ethics Committee of Hospital Israelita Albert Einstein (11) 2151-3729) and the Customer Service (SAC) (11) 2151-0222 any question that has to do with this study or about my rights as a participant.
- 2. My participation in this research study is strictly voluntary. I can refuse to take part in this study without any penalty or loss of benefits to which I am entitled. I can also withdraw from the study at any time without any penalty or loss of my rights. If you withdraw your authorization, you will be removed from the study and the Principal Investigator and staff will no longer use or disclose your information.
- 3. I understand that the study can be modified or stopped at any time by the Principal Investigator or the Ethics Committee of Hospital Israelita Albert Einstein. If this occurs, I will be informed immediately.
- 4. I will be informed of any new findings that may affect my willingness to continue being part of the study.
- 5. The Principal Investigator and Hospital Israelita Albert Einstein will take appropriate steps to keep my personal information private. However, there is no guarantee of absolute privacy. Federal agencies such as ANVISA and the Ethics Committee of Hospital Israelita Albert Einstein, can review my records to collect data or to check if the research is being done safely and correctly.
- 6. I understand that there are no plans to compensate me for any patents or discoveries that may result from my participation in this research. I will not receive compensation for participating in this study. No amount will be refunded for my participation in this survey.


| Researcher Rubric | Participant rubric |
|--------------------------|--------------------|
| Version 2 - January 2020 | |



7. Having read and understood the information above and having the opportunity to ask questions about this study, think about the study, and speak with others when necessary, I give permission to the Principal Investigator to register for that study. By signing this consent form, I am not giving up any of my legal rights. I was provided with a signed copy of that consent document and all blanks were filled.

| Full | name of the | e researc | h participant | | |
|---|---|---|---|---|---|
| Si | gnature of ı | research | Date:<br>participant | I | _/ |
| Full and legible nam | e of the per | son respo | onsible for obt | aining | consen |
| Signature of th | ne person re | sponsibl | Date:_<br>e for obtaining | | |
| Oignature of th | ie person re | оронова | | , 001130 | Jiit. |

|----------|
|----------|



## Informed Consent Form (ICF) - NURSE

Researchers: Prof. Dra Eliseth Ribeiro Leão (Advisor) Enfa Lidiane Soares Sodré da Costa (Master Degree Student)

# Research title: "Evidence-Based Practice: Proposed Application of Facilitating Tools for Clinical Nurses"

Dear nurse:

Version 2 - January 2020

We would like to invite you to participate as a volunteer in the research entitled: "Evidence-Based Practice: Proposal for the Application of Facilitating Tools for Clinical Nurses", which refers to the Professional Master's Course Completion Course Teaching in Health. The objectives of this study are:

- 1) Verify the adequacy of the authorized translation of the Portuguese language version of the guide tools of the Johns Hopkins Center for Evidence-Based Practice (Johns Hopkins Center for Evidence-Based Practice), located in the United States.
- 2) Analyze, from the perspective of the clinical nurse, whether these tools are facilitators in structuring and describing an evidence-based practice project (EBP);
- 3) Analyze, from the researcher's perspective, whether the PBE project met the requirements of: elaboration of a clinical question, bibliographic survey, critical evaluation of the evidence, summary of the evidence and elaboration of the dissemination plan;
- 4) Verify whether previous attitudes and knowledge regarding the implementation of PBE influence the structuring of a PBE project.

His form of participation in the study consists of initially answering the questionnaire: Evidence-Based Practice and Clinical Effectiveness EBPQ, this instrument assesses attitudes and knowledge about Evidence-Based Practice (EBP). Afterwards, he will participate in a six-hour workshop on PBE, divided into two days that will include content and practical class.

The participation of the workshop will be conducted as follows: we will divide the participants into 2 groups, the determination of which group you will participate in will be carried out at random, through a draw, neither the

|-------------------|----------------------|
| Researcher Rubric | _ Participant rubric |



participant nor the researcher being able to decide in which group you will participate.

Group A): will receive theoretical and practical training in PBE through a structured model workshop with themes related to the introduction to PBE, formulation of a practical question, bibliographic survey to search for evidence, critical analysis of evidence, classification of level and quality of evidence, summary and dissemination plan, with the final proposal of a practical class that aims to structure and describe an individual case through an exercise designed to go through the phases of a PBE project, as the basis for this exercise we will use a finalized and consolidated project, this will be used as a template for the exercise.

Group B): will receive the same training as Group A, plus the presentation and availability of the guide tools of the Johns Hopkins Center for Evidence-Based Practice in Portuguese to be used in the practical class for the structuring and individual description of the PBE exercise case, each tool has a brief description of the content of how to fill it out. The same theme of the case will be used in both groups.

We ask that at the end of the workshop answer a second questionnaire: Structural Assessment Questionnaire and description of an EBP project from the perspective of the Nurse, this questionnaire aims to assess how much the content offered in the workshop was facilitating for you in the structuring and description of a PBE project. This questionnaire should take an average of five minutes to complete.

The questionnaires will be inserted in the REDcap® digital platform, you will have access to electronic resources notebook or tablet to insert your answers.


| Researcher Rubric | Participant rubric _ |
|-------------------|----------------------|



You will receive follow-up from the researcher during the workshops and the content produced in the practical class will be evaluated through a third questionnaire to be completed by the researcher: Compliance verification questionnaire in the exercise of preparing a PBE project from the researcher's perspective

You will not be charged anything and you will not be charged for your participation in this survey. The project envisages that the workshops take place during working hours, without the need for costs associated with transportation or food.

Regarding the risks of your participation in this research, the form may contain questions that need clarification with minimal risk of wear and tear. You can refuse to answer any questions that make you feel uncomfortable. If you have concerns after completing the form, you are encouraged to contact the person responsible for the study.

In addition, only researchers will have access to personal information and data. To minimize the risk of exposure and guarantee its anonymity, the researchers commit to not using your name or any other data that can identify you at any stage of the research. There are no other risks related to your participation in the project.

There is an expected benefit for you, if you participate in this project with regard to deepening the theme of practice based on evidence and use of this knowledge acquired during the exercise of your profession.

We emphasize that your participation in this research is independent of your professional or academic activity at the institution, it is ensured that there will be no type of retaliation if you refuse to participate in this research.

|-------------------|--------------------|
| Researcher Rubric | Participant rubric |

Version 2 - January 2020



#### I understand that the following statements about this research are true:

I can ask any question to the person in charge of the study, Lidiane Soares Sodré da Costa. I can contact you at (11) 99625-3924. I can also contact the Ethics Committee of the institution (Research Ethics Committee of Hospital Israelita Albert Einstein (11) 2151-3729 and the Customer Service (SAC) (11) 2151-0222 any question that has to do with this study or my rights as a participant.

- 1. My participation in this research study is strictly voluntary. I can refuse to take part in this study without any penalty or loss of benefits to which I am entitled. I can also withdraw from the study at any time without any penalty or loss of my rights. If you withdraw your authorization, you will be removed from the study and the Principal Investigator and staff will no longer use or disclose your information.
- 2. I understand that the study can be modified or stopped at any time by the Principal Investigator or the Ethics Committee of Hospital Israelita Albert Einstein. If this occurs, I will be informed immediately.
- 3. I will be informed of any new findings that may affect my willingness to continue being part of the study.
- 4. The Principal Investigator and Hospital Israelita Albert Einstein will take appropriate steps to keep my personal information private. However, there is no guarantee of absolute privacy. Federal agencies, such as ANVISA and the Ethics Committee of Hospital Israelita Albert Einstein, can review my records to collect data or to check if the research is being done safely and correctly.
- 5. I understand that there are no plans to compensate me for any patents or discoveries that may result from my participation in this research. I will not receive compensation for participating in this study. No amount will be refunded for my participation in this survey.


| Researcher Rubric | Participant rubric |
|-------------------|--------------------|

Version 2 - January 2020



- 6. Having read and understood the information above, and had the opportunity to ask questions about this study, think about the study, and speak to others when necessary, I give permission to the Principal Investigator to register for that study.
- 7. By signing this consent form, I am not giving up any of my legal rights. I was provided with a signed copy of that consent document and all blanks were filled.

| Full name of the research participant |
|----------------------------------------------------------------------|
| Date://<br>Signature of research participant |
| Full and legible name of the person responsible for obtaining conser |
| Date://<br>Signature of the person responsible for obtaining consent |
| Signature of the person responsible for obtaining consent |
| Page |

Researcher Rubric \_\_\_\_\_\_ Participant rubric \_\_\_\_\_